CLINICAL TRIAL: NCT00137514
Title: Chloroquine and Amodiaquine for Treatment of Symptomatic Children With Plasmodium Malaria in Guinea-Bissau
Brief Title: Chloroquine and Amodiaquine for Treatment of Malaria in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSB-2001-chl-amo; 2004-126 (SAREC).
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Malaria, Falciparum
Keywords: malaria; Plasmodium falciparum; chloroquine; amodiaquine; treatment; Guinea-Bissau; children
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Chloroquine; Amodiaquine

INTERVENTIONS:
Drug: chloroquine
Drug: amodiaquine

SUMMARY:
This study will evaluate the efficacy of the treatment recommended by the National Malaria Programme in Guinea-Bissau as compared to a higher dose of chloroquine and to another anti-malarial drug, amodiaquine. The genetic basis of the parasites for developing resistance will be examined. Children coming to Bandim Health Centre with symptoms of malaria and a positive malaria test will be included. The children will be visited and malaria films will be obtained weekly until day 35. In case of a reappearance of parasites the children will be re-treated with sulfadoxine/pyrimethamine.

DETAILED DESCRIPTION:
This study compares treatment of uncomplicated malaria in children in Guinea-Bissau as recommended by the national malaria programme (chloroquine in a total dose of 25 mg/kg), either with a total dose of 50 mg/kg chloroquine or with a total dose of 15 or 30 mg of amodiaquine. As both annual in vitro studies (from 1992 to 2004 except 1998, 1999) and several in-vivo studies from Guinea-Bissau indicate a fairly stable chloroquine resistance prevalence, another aim of this study is to evaluate the genetic basis of chloroquine resistance in Guinea-Bissau by analyzing specific single nucleotide polymorphisms in pfcrt and pfmdr1 in blood samples from this in vivo trial.

Following consent to participate, children visiting the Bandim Health Centre on the outskirts of Bissau with mono-infection with Plasmodium falciparum are by block-randomization allocated to one of the four different treatment groups. The treatment is given supervised by one of the health workers. The children are visited and malaria films obtained on day 2 and day 7 and then once weekly until day 35. On day seven, 100 microliters of capillary blood are drawn for analyses of chloroquine or amodiaquine concentrations in whole blood. Whenever a child has recurrent parasitaemia, a filter-paper blood-sample is collected for later PCR analysis.

If parasites reappear in 50% or more of at least 40 children in one of the treatment groups this treatment arm should be terminated. During the study parents are recommended to bring the child to Bandim Health Centre in case of any illness. Participating children will be examined and treated free of charge. Following the recommendations of the national Malaria Programme sulfadoxine/pyrimethamine will be used for re-treatment of children in case of recrudescence.

The results from this study could be used when giving the needed new recommendations for treatment of malaria in Guinea-Bissau. If still effective mono-therapy with a higher dose of chloroquine could be used until the introduction of a better treatment is possible. When artemisinine combination therapy is going to be introduced in Guinea-Bissau the results could be helpful in deciding if amodiaquine should be considered as the partner drug - and in which dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 15 years of age presenting at Bandim Health Centre
* Symptoms suggestive of malaria
* At least 20 P. falciparum parasites per 200 leukocytes in a thick film
* Live in Bandim (to enable follow-up)

Exclusion Criteria:

* Severely ill children considered needing the services of a hospital by the medical doctor in charge
* Stated medication with other antimalarials within one week prior to treatment
* Previous idiosyncratic reactions to any of the study drugs

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720
Dates: Start 2001-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Parasite reappearance rate
hospitalization during follow-up

SECONDARY OUTCOMES:
Genetic markers in parasites
recrudescence rate
re-infection rate

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau Region, Guinea-Bissau

REFERENCES:
- [Derived] Jovel IT, Kofoed PE, Rombo L, Rodrigues A, Ursing J. Temporal and seasonal changes of genetic polymorphisms associated with altered drug susceptibility to chloroquine, lumefantrine, and quinine in Guinea-Bissau between 2003 and 2012. Antimicrob Agents Chemother. 2015 Feb;59(2):872-9. doi: 10.1128/AAC.03554-14. Epub 2014 Nov 24. PMID 25421474